CLINICAL TRIAL: NCT04005677
Title: The Early Diagnosis of Pulmonary Nodule Based on Multi-dimension Messages
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: Whuh2019 v.1
Record Dates: First submitted 2019-06-23; First posted 2019-07-02 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Nodule, Solitary; Lung; Node
MeSH Terms: conditions — Solitary Pulmonary Nodule | interventions — Urination; Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- lung cancer
  Interventions: Diagnostic Test: The serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics are collected.
- benign lung nodule
  Interventions: Diagnostic Test: The serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics are collected.
- lung nodule
  Interventions: Diagnostic Test: The serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics are collected.

INTERVENTIONS:
Diagnostic Test: The serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics are collected. — The serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics including age, sex, smoking status, BMI, address, greening environment and the laboratory tests are collected to to analyze the ctDNA, RNA, protein, metabolites, immune status and their relationships with the tumorigenesis and the gene mutation of lung cancer.

SUMMARY:
The researchers are aimed to investigate the early diagnosis of pulmonary nodule based on DNA, RNA, protein, metabolites through analyzing the serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and clinical characteristics.

DETAILED DESCRIPTION:
By recruiting people with pulmonary nodules identified by CT scans, three groups are confirmed as the lung cancer group, the benign lung nodule group who are identified by pathological analysis, and the small lung nodule group that should be followed up. Then the serum, plasma, urine, faeces, peripheral blood mononuclear cell (PBMC), exhaled breath condensate and the clinical characteristics including age, sex, smoking status, BMI, address, greening environment and the laboratory tests are collected to analyze the ctDNA, RNA, protein, metabolites, immune status and their relationships with the tumorigenesis and the gene mutation of lung cancer.

ELIGIBILITY:
Inclusion Criteria:

For lung cancer groups

* (1) Patients diagnosed with lung cancer;
* (2) Clear diagnosis by pathological examination to determine pathological type;
* (3) Those aged 18-80 years old;
* (4) For patients with newly diagnosed lung cancer, CT confirmed that the size of primary lung cancer is ≤ 3 cm;
* (5) The patient or family member agrees to participate in the study and sign an informed consent form;
* (6) No other serious cardiopulmonary diseases. For lung nodule
* (1) Those aged 18-80 years;
* (2) CT clear lung nodule size ≤ 3cm;
* (3) 1-3cm pulmonary nodules confirmed by pathological diagnosis as non-lung cancer or other metastatic cancer patients or ≤1cm pulmonary nodules
* (4) The patient or family member agrees to participate in the study and sign an informed consent form;
* (5) No other serious cardiopulmonary diseases.

Exclusion Criteria:

* (1) Women who are breast-feeding, pregnant or preparing for pregnancy;
* (2) Those who are allergic to allergies and multiple drugs;
* (3) Combining severe primary diseases such as cardiovascular and cerebrovascular, liver, kidney, and hematopoietic system, as well as subjects with mental illness;
* (4) concurrently infected;
* (5) Those who participated in other clinical trials within three months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled are volenteered and are willing to be followed up.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Up-regulation of ctDNA | the first day subjects are enrolled the outcome will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China